CLINICAL TRIAL: NCT01902511
Title: A Trial to Study the Influence of Growth Factors on Bone Marrow and Hepatic Regeneration in Patients With Decompensated Cirrhosis.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ILBS-Hepatic Regeneration -001
Record Dates: First submitted 2013-07-15; First posted 2013-07-18 (Estimated); Last update posted 2016-11-22 (Estimated); Status verified 2016-02

CONDITIONS: Decompensated Cirrhosis
MeSH Terms: interventions — Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- G-CSF + Erythropoietin (Experimental)
  Interventions: Drug: G-CSF
- G-CSF (Active Comparator)
  Interventions: Drug: G-CSF+Erythropoetin

INTERVENTIONS:
Drug: G-CSF+Erythropoetin
  Arms: G-CSF
Drug: G-CSF
  Arms: G-CSF + Erythropoietin

SUMMARY:
This will be a randomized double blind study which will be conducted on patients admitted to Department of Hepatology from June 2013 to may 2014 at ILBS, New Delhi. Patients not having any exclusion criteria will undergo bone marrow examination and liver biopsy at the baseline.

60 patients of decompensated cirrhosis will be randomised into two limbs- limb A (30 patients) will receive G-CSF and erythropoietin while those on limb B (30 patients) will receive G-CSF alone. The drugs will be given for 2 months and patient will be followed for 1 year. G-CSF will be given at a dose of 5 µg/kg s/c at days 1, 2, 3, 4, 5 and then every 3rd day till day 60 (total 22 doses). Erythropoietin will be given s/c at dose of 500 IU/Kg twice a week for 2 months.

Follow up will be done on days 0,3,7,14,28, day 42 (6 weeks), day 60 (2 months), day 90 (3 months), day 180 (6 months), day 270 (9 months); and day 360 (1 year).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18-65 years
* All patients who are known to have cirrhosis of liver with portal hypertension and are compensated on presentation with no features of ascites/ jaundice/ bleed/ HE/ HRS.
* Only patients with alcoholic cirrhosis and cryptogenic cirrhosis (etiology work up negative) will be enrolled in the study.

Exclusion Criteria:

* Sepsis ( Any culture positive: blood, urine, any other obvious source of infection: UTI, LRTI)
* Variceal bleed in the past 3 months
* Autoimmune disorders
* HCC (Hepatocellular Carcinoma)
* Multi organ failure
* Any features of decompensation in form of ascites/Jaundice/ HE (grade 3 or 4) / HRS
* HIV seropositivity
* Essential hypertension
* Pregnancy
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2013-07; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
The primary end point will be transplant free survival rate at 1 year in patients with decompensated cirrhosis. | 1 Year

SECONDARY OUTCOMES:
Histopathological evidence of hepatic regeneration and mobilization of CD34/stem cells | 1 Year
Histopathological evidence of contribution of bone marrow precursor cells in hepatic regeneration and the markers predicting positive response to growth factors | 1 Year
Development of new complications such as appearance or worsening of hepatic encephalopathy, hepatorenal syndrome and sepsis. | 1 Year
Improvement in severity assessment scores and safety profile of G-CSF (Growth-Colony Stimulating Factor) + EPO (Erythropoetin)dual therapy vs. G-CSF alone. | 1 Year
Transplant free survival at 6 months in both groups | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Dr Lovkesh Anand, MD, Principal Investigator — Institute of Liver & Biliary Sciences.
Locations (1):
- Institute of Liver & Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Kumar D, Maheshwari D, Nautiyal N, Shubham S, Rooge S, Anand L, Vyas A, Kumari R, Sharma S, Bihari C, Mohanty S, Maiwall R, Kumar A, Sarin SK. Defects in energy metabolism are associated with functional exhaustion of bone marrow mesenchymal stem cells in cirrhosis. Am J Stem Cells. 2022 Feb 15;11(1):12-27. eCollection 2022. PMID 35295591
- [Derived] Anand L, Bihari C, Kedarisetty CK, Rooge SB, Kumar D, Shubham S, Kumar G, Sahney A, Sharma MK, Maiwall R, Kumar A, Sarin SK. Early cirrhosis and a preserved bone marrow niche favour regenerative response to growth factors in decompensated cirrhosis. Liver Int. 2019 Jan;39(1):115-126. doi: 10.1111/liv.13923. Epub 2018 Aug 10. PMID 29962032